CLINICAL TRIAL: NCT05957861
Title: Exploring the Effectiveness and Trajectory of Adherence to Web-based Exercise Among Community-dwelling Adults With High Body Fat
Brief Title: Exploring the Effectiveness to Web-based Exercise Among Community-dwelling Adults With High Body Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Tainan Junior College of Nursing (Other)
Responsible Party: Principal Investigator, Yu-Hsuan Chang, Assistant professor, National Tainan Junior College of Nursing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: National Tainan Junior College
Record Dates: First submitted 2023-06-28; First posted 2023-07-24 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Adherence, Treatment; Exercise
Keywords: web-based exercise; adherence; body composition
MeSH Terms: conditions — Treatment Adherence and Compliance; Motor Activity

STUDY DESIGN:
Intervention Model Description: we will design a randomized controlled trial comprising two arms of a 16-week exercise web-based aerobic exercise (AE) training and another control group without any exercise intervention.
Who Masked: Outcomes Assessor
Masking Description: PI will be blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- web-based exercise (Experimental): Participants will receive web-based aerobic exercise (AE) training three times per week for 16 weeks.
  Interventions: Behavioral: web-based aerobic exercise
- control group (No Intervention): control group without any intervention.

INTERVENTIONS:
Behavioral: web-based aerobic exercise — Our designed AE program involved core muscle training through movements including marching, step touches, lunges, v-steps, box steps, twists, knee-ups, scoops, and scissors.
  Arms: web-based exercise

SUMMARY:
The study findings can derive an effective exercise type either web-based or supervise exercise as well as build a series of exercise video that can promote self-exercise at home for health promotion for community residents.

DETAILED DESCRIPTION:
Background: Web-based exercise is effective alternative training for community residents on health improvement; however, adherence to their performance is challenging.

Purpose: This study aimed to (1) compare the effectiveness of 16-week exercise on improving blood samples, body composition, and anthropometric parameters between web-based exercise and supervised exercise; and (2) examine the trajectory of exercise adherence of web-based exercise for attendance and intensity over time for community-dwelling adults with high body fat.

Design: A two-arm randomized control trial. Method: Participants who received 16-week supervised exercise for aerobic exercise training on 2020 in our previous project was served as one of control groups (n = 34). In present project, purposive sampling will be used to enroll a target of 66 community-dwelling residents aged 40-64 years with inactive habits and body fat percentage ≧ of 25% for males and ≧ 30% for females in study. Eligible participants will be stratified by sex and then block randomly divided into web-based exercise or a control group (without any exercise intervention). The web-based exercise will prescribe a 30-minute of aerobic exercise at least moderate intensity prescription for three times per week. Heart rate reserve and self-perceived exertion will be self-recorded on the web by participants. Generalized estimating equations will be used to explore the effectiveness of web-based exercise.

Implications: The study findings can derive an effective exercise type either web-based or supervise exercise as well as build a series of exercise video that can promote self-exercise at home for health promotion for community residents.

ELIGIBILITY:
Inclusion Criteria:

* aged from 40 to 64 years.
* have a body fat percentage of ≧25% if a man or ≧30% if a woman.
* can use the internet for watching the exercise video online.
* with inactive habit (≤ 3 days of physical activity per week and ≤ 30 min per session).

Exclusion Criteria:

* blind.
* currently under diet control.
* with any unsafety concern for their condition, such as pregnancy, myocardial infarction, stroke, or body fat percentage of ≧40%.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
The change of cholesterol | two times (from baseline to the end of 16-week)
  the unit is mg/dl
The change of fasting sugar from blood sample | two times (from baseline to the end of 16-week)
  the unit is mg/dl
The change of insulin from blood sample | two times (from baseline to the end of 16-week)
  the unit is μIU/mL
The change of weight | two times (from baseline to the end of 16-week)
  weight in kilograms, will be measured using body composition analyzer
The change of waist circumference | two times (from baseline to the end of 16-week)
  the unit is centimeters
The change of body fat percentage | two times (from baseline to the end of 16-week)
  the unit is %, will be measured using body composition analyzer
The change of visceral fat | two times (from baseline to the end of 16-week)
  the unit is square centimeters, will be measured using body composition analyzer
The change of hip circumference | two times (from baseline to the end of 16-week)
  the unit is centimeters.
The change of High-density lipoprotein [HDL] | two times (from baseline to the end of 16-week)
  the unit is mg/dl
The change of low-density lipoprotein [LDH] | two times (from baseline to the end of 16-week)
  the unit is mg/dl
The change of triglycerides [TG] | two times (from baseline to the end of 16-week)
  the unit is mg/dl

SECONDARY OUTCOMES:
Adherence measurement | Each exercise session
  Number of sessions attended/ Number of total sessions prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsuan Chang, phD, Principal Investigator — National Tainan Junior College of Nursing

IPD SHARING:
Plan to Share IPD: No
for research privacy.